CLINICAL TRIAL: NCT03230240
Title: Immunologic, Cellular, and Anti-microbial Profiling of Intraperitoneal Chemotherapy
Brief Title: Immunologic Profile of Peritoneal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MercyOne Des Moines Medical Center (Other)
Responsible Party: Principal Investigator, Jan Franko, MD, Surgical Oncologist, MercyOne Des Moines Medical Center
Other Study IDs: MMC2015-62
Record Dates: First submitted 2016-02-08; First posted 2017-07-26 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Carcinomatosis
MeSH Terms: conditions — Carcinoma | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — ascites
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIPEC: Patients with carcinomatosis or other peritoneal surface malignancy
  Interventions: Drug: HIPEC

INTERVENTIONS:
Drug: HIPEC — heated intraIP chemotherapy
  Other Names: Hyperthermic intraperitoneal chemotherapy

SUMMARY:
To ascertain immunologic profile of peritoneal cavity and its relationship to immediate postsurgical outcome (morbidity or the treatment) and long-term outcome (time to recurrence and survival).

DETAILED DESCRIPTION:
1. BACKGROUND:

   Tumor-host interaction includes inactivation of immunologic recognition of malignant cells by a mechanism yet not fully understood. Aneuplodity studies on cells from different metastatic sites demonstrate increased heterogeneity depending on metastatic site (Kimball 1997). This suggests that phenotypically different cell populations are responsible for different metastases and may demonstrate different sensitivity/resistance to treatment. Kitayama (2015) studied ratio of lymphocytes to epithelial cell in peritoneal cavity, but used this ratio only as marker of tumor burden and did not relate it to perioperative outcome.

   Investigators have clinically observed a different behavior of peritoneal metastases as compared to those located in other body sites (Franko 2012, Klaver 2012, Franko 2016). It is hypothesized that tumor-host interaction and host-treatment response are related to treatment-related morbidity, early vs. delayed recurrence, and overall survival.

   There is a limited literature and research examining the immunologic profile of intraperitoneal chemotherapy and its relationship to morbidity and future metastatic sites. Therefore, further knowledge of the biology of different peritoneal surface metastatic disease is necessary. This, with additional research, may lead to specific therapies.
2. OBJECTIVES:

   To ascertain immunologic profile of peritoneal cavity and its relationship to immediate postsurgical outcome (morbidity or the treatment) and long-term outcome (time to recurrence and survival).
3. STUDY POPULATION:

   Patients with peritoneal carcinomatosis undergoing intraperitoneal chemotherapy.

   3.1 Exclusion criteria: Under age of 18 years, pregnant patients, those unable to provide consent.
4. SUBJECT RECRUITMENT METHODS:

   All patients scheduled to undergo cytoreductive procedure for peritoneal carcinomatosis in at Mercy Medical Center in Des Moines, IA (MMC). This study will be offered during a preoperative office or a hospital visit by Dr Franko or Dr Goldman.
5. INFORMED CONSENT:

   Attached
6. RESEARCH PROCEDURES:

   Liquid samples will be collected and analyzed. We will collect ascites, peritoneal washout, HIPEC perfusion fluid. Samples will be analyzed using flow cytometry, routine fluid cytology, and tested for anti-microbial properties.

   6.1 Sample labeling:

   The following peritoneal fluid sample will be collected:

   A - ascites or peritoneal saline washout at the beginning of case B - HIPEC fluid after pre-heating and immediately before chemotherapy agent provision C, D, E - HIPEC fluid at 30, 60, and 90 minutes of perfusion 6.2 Flow cytometry Fluid samples will be run through flow cytometry to analyze proportion of CD3, CD4, CD8, CD20, CD34 positive cells.

   6.3 Cytology Routine cytology of peritoneal fluid represents standard of care for malignant disease diagnostics and will be conducted as per usual diagnostic plan.

   6.4 Detection of anti-microbial properties Fluid samples will be introduced to bacterial growth in the microbiology laboratory at MMC. Growth inhibition of standard bacterial strains (Staphylococcus aureus, Escherichia coli) will be recorded. The samples will also be sent for flow cytology and possibly chromatography to measure exact concentrations of chemotherapeutic agent remaining in samples.

   6.5 High-performance liquid chromatography A limited number of samples will be analyzed with high performance liquid chromatography to determine exact chemotherapy concentration remaining in sample (den Hartigh 1981). This part of the research is conducted in collaboration with Dr. Brian Gentry at Drake University. Sample provided for this part of research will be deidentified, date-time-stamped, and Drake's team will receive no other clinical or demographic information. Re-identification at MMC remains possible.

   To satisfy methodological needs, we will collect each case will provide 2 samples: Sample B will be a HIPEC perfusate solution at the completion of initial heating up period collected before adding chemotherapy agent. Sample E will be perfusate at the completion of HIPEC procedure expected to contain MMC. Sample E is the main research sample. Sample volume is 5 cc.
7. DATA COLLECTION AND ANALYSIS:

   Sample B is obtained before active treatment agent is provided to the solution. It represents a small withdrawal volume of 5 cc out of approximately 3-5 liter HIPEC solution used in usual case. Average clinical dosing of carrier solution is 2 liters/m2 of patient's body surface area, therefore representing < 0.2% total HIPEC carrier solution volume. Sample C & D represent the same volume, but are withdrawn from patient with active treatment. Given very small volume of each sample no negative effect is expected, as total sample volume is <0.6% total HIPEC perfusion fluid.

   All other research samples are derived only from residual surgical specimen exclusively obtained for treatment purposes. Data collection will include, but is not limited to, patient name, gender, age, initial tumor stage, current tumor stage & extent, histology, prior treatment modalities, and results from flow cytometry, microbiology, and HPLC, and medical record for 60 months following surgery.
8. POTENTIAL RISKS:

   8.1 Risks related to sampling: Some body fluid samples are collected on residual surgical specimens removed from patient for treatment purpose (samples A and E), and are independent of research. The exception are Sample B,C,D - the only samples removed from patient for research purpose only. The volume of each sample is minute, < 0.2% of total perfusate volume; therefore total sampling volume in ≤0.6% expected perfusate volume. Given these two facts it is reasonable to assume no expected influence on patients' outcome.

   8.2 Risks related to loss of confidentiality Because identifiable data are collected there is a potential risk of breach of confidentiality. To protect confidentiality and minimize risk, research data will be maintained on MMC computers with access restricted to the core research team and password-protected file. Privacy laws will be maintained.
9. RESEARCH MATERIALS, RECORDS, AND PRIVACY:

   Research database will be maintained on MMC computers with privileged access restricted to the core research team and password-protected file. Privacy laws will be maintained.
10. CONFIDENTIALITY:

No research specimen will be stored. All research specimens will be destroyed in accordance with usual laboratory procedures.

Electronic data will be maintained until the last analysis is carried out. Access to the data will be limited to authorized personnel associated with this study.

The samples provided to Drake University are deidentified and cannot be re-identified by Drake University team. Therefore no confidentiality loss there is expected.

ELIGIBILITY:
Inclusion Criteria:

* HIPEC pt

Exclusion Criteria:

* absent consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peritoneal carcinomatosis undergoing intraperitoneal chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
In vitro growth of Staph Aureus and Escherichia coli measured in millimeters of colony forming unit on Agar plate | 1 year after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jan Franko, MD, PhD, Principal Investigator — MercyOne Des Moines Medical Center
Locations (1):
- MercyOne Des Moines Medical Center, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Franko J, Brahmbhatt R, Tee M, Raman S, Ferrel B, Gorvet M, Andres M. Cellular Immunoprofile of Peritoneal Environment During a HIPEC Procedure. Ann Surg Oncol. 2020 Dec;27(13):5005-5013. doi: 10.1245/s10434-020-08870-3. Epub 2020 Jul 21. PMID 32696309